CLINICAL TRIAL: NCT01021449
Title: Epigenetic Regulation of BDNF and TrK B in Schizophrenic Patients
Brief Title: Epigenetic Regulation of BDNF in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tiao-Lai Huang, Head of Department of Psychiatry, Chang Gung Memorial Hospital
Other Study IDs: CMRPG870951 and CMRPG870952
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: BDNF, DNA Methylation, Suicide, Drug Responses.
Keywords: schizophrenia, BDNF, DNA methylation, histone modification
MeSH Terms: conditions — Suicide; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Healthy subjects
- Schizophrenia: Schizophrenic patients

SUMMARY:
In this proposal, we will (1) detect the associations between BDNF and Trk B gene DNA methylation, histone modification, psychotic symptoms, obesity, suicide and antipsychotic drug responses in Taiwanese patients (2) discuss the possible mechanisms of epigenetic regulation of BDNF and Trk B in schizophrenia patients.

DETAILED DESCRIPTION:
A total 160 subjects (80 subjects every year, including 40 healthy controls and 40 schizophrenia patients) will be recruited during a 2-year period. The first year, the baseline data of BDNF and Trk B DNA methylation, protein and mRNA levels in all subjects will be collected and the following 1 months data will also be collected in schizophrenia with antipsychotic drug treatments. The second year, the baseline data of BDNF and Trk B histone modification in all subjects will be collected.

ELIGIBILITY:
Inclusion Criteria:

-

1. The clinical screening and assessment in schizophrenic patients：

1. 40 schizophrenia patients will be recruited in psychiatric inpatients according to DSM-IV criteria (APA, 1994) by a structured interview (SCID). The assessment will be done by two senior psychiatrists. The intra-rater and inter-rater reliability will be done before this project started
2. age : 18-65 years old.
3. The patients had the ability to complete the written inform consent.。
4. The choice of antipsychotic drugs depended on the need of patients in natural treatment procedure. They included conventional drugs, eg.haloperidol 10-20 mg/day；SDA (serotonin dopamine antagonist) drug, eg. clozapine 100-400 mg/day or risperidone 3-6mg/day. The choice of the medication was according to the need of patients including previous responses and side effects.
5. PANSS (Positive and Negative Syndrome)(Kay, 1987,1988&1989) for positive, negative symptoms and severity.
6. Check body mass index (BMI): if BMI<24: normal; 24<BMI<27: overweight; BMI>27: obesity (Taiwan criteria, 2004). If the patients were overweight or obesity, the lipid profiles would be done and we would consult the experts to assess these patients. The condition for diet control and daily activity will be observed. If the condition was extremely abnormal, the case will be excluded.
7. Suicide behavior in tis study includes complete suicide and suicide attempt.

Exclusion Criteria:

1. The patients had systemic diseases, including metabolic, heart, and liver diseases。
2. The patients had received any drugs before entering this protocol.
3. The patients were heavy smokers or dependent on alcohol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in our clinical setting. By a semi-structured interview for DSM-IV criteria, total 160 subjectes (80 subjects every year, including 40 healthy controls and 40 schizophrenia patients with acute exacerbation) will be recurited during a 2-year period. The data of blood BDNF and Trk B DNA methylation and histone remodelling of all subjects will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
BDNF and Trk B DNA methylation, protein and mRNA levels | Two years

SECONDARY OUTCOMES:
the associations between BDNF and Trk B gene DNA methylation, histone modification, psychotic symptoms, obesity, suicide and antipsychotic drug responses in Taiwanese patients | two years

CONTACTS AND LOCATIONS:
Overall Officials: Tiao-Lai Huang, M.D., Principal Investigator — Chang-Gung Memorial Hospital, Kaohsiung
Locations (1):
- Department of Psychiatry, Chang Gung Memorial Hospital, Kaohsiung City, Taiwan